CLINICAL TRIAL: NCT05495243
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of ARINA-1 in Adult Participants With Non-cystic Fibrosis Bronchiectasis (NCFBE) With Excess Mucus and Cough
Brief Title: Phase 2a, 28-day Investigational Use Study of ARINA-1 in Non-Cystic Fibrosis Bronchiectasis (NCFBE) With Excess Mucus and Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVN-301
Record Dates: First submitted 2022-06-24; First posted 2022-08-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARINA-1 (Experimental): ARINA-1 (88 mg/mL ascorbic acid, ASC; 150 mg/mL reduced glutathione, GSH); fixed dose, 4 mL solution inhaled twice daily via nebulization for 28 days
  Interventions: Drug: ARINA-1
- Placebo (Placebo Comparator): Isotonic saline (0.9%); 4 mL solution inhaled twice daily via nebulization for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARINA-1 — ARINA-1 (88 mg/mL ascorbic acid, ASC; 150 mg/mL reduced glutathione, GSH)
  Arms: ARINA-1
Drug: Placebo — Isotonic saline (0.9%)
  Arms: Placebo

SUMMARY:
This is a randomized, Phase 2a, double-blind, placebo-controlled study to evaluate the safety and efficacy of ARINA-1 compared to placebo (isotonic saline, 0.9%) in participants with NCFBE. Study participants will receive either study treatment or placebo twice daily for 28 days. Efficacy endpoints will include quality of life, sputum rheological markers, and blood inflammatory markers. Quality of life will be measured using the following tools: Quality of Life-Bronchiectasis (QOL-B) questionnaire, St. George's Respiratory Questionnaire (SGRQ), Chronic Airways Assessment Test (CAAT), and a daily clinical global impression questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NCFBE confirmed by chest CT
* 18-80 years old, inclusive at time of informed consent
* BMI >18
* Percent predicted FEV1 > 40%, pre-bronchodilator
* Stable for 90 days with any airway clearance technique (ACT) method(s)
* Stable on standard of care (SOC) therapy for 90 days (includes cycling antibiotics, such as inhaled tobramycin, and long-term macrolide therapy) and not likely, in the opinion of the investigator, to require any changes to therapy during the duration of study participation
* Fully vaccinated for COVID-19 (second dose of a 2-shot regimen or single dose of 1-shot regimen completed >14 days prior to the screening visit)
* Must be able to produce a sputum sample
* If female and of childbearing potential, must be willing to use contraception for the duration of the study.

Exclusion Criteria

* Positive urine pregnancy test for women of childbearing potential (WOCBP) at screening and baseline visit
* Active exacerbation ≤28 days prior to the baseline visit
* Initiating or changing antibiotic, antiviral, or antifungal therapy ≤ 28 days prior to the baseline visit
* Changing or initiating any vitamin C, glutathione or N-acetyl-cysteine-containing therapy or multivitamin within 30 says prior to the screening visit.
* Positive COVID-19 diagnostic test (PCR or antigen) within 90 days prior to the screening visit.
* Participated in other interventional drug or device studies within 30 days of the screening visit (Note: observational studies are acceptable)
* Significant unstable comorbidities (in the opinion of the site investigator), such as heart failure, cardiovascular disease, diabetes, renal disease, liver disease
* Current tobacco or marijuana smoker (those with active smoking exposure <180 days prior to the screening visit) (Note: edibles are acceptable)
* Requiring the use of any supplemental oxygen
* Currently on cycled antibiotics (e.g., tobramycin) or have been on a cycled antibiotic regimen within 90 days prior to the screening visit.
* Current diagnosis of non-tuberculous mycobacteria (NTM) requiring antibiotic treatment. (Participants who test positive for NTM but who are not currently on antibiotic therapy are eligible for screening)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 56 days
  Incidence of participants that experience an adverse event following administration of treatment
Proportion of participants that experience each treatment-emergent adverse event | 56 days

SECONDARY OUTCOMES:
Compare quality of life (as measured by CAAT questionnaire) between the ARINA-1 and placebo arms | 56 days
  8 questions rated on a 0-5 scale
Compare quality of life (as measured by SGRQ) between the ARINA-1 and placebo arms | 56 days
  42 questions, ranked on a 5-point descriptive scale or true/false
Compare quality of life (as measured by QOL-B) between the ARINA-1 and placebo arms | 56 days
  37 questions ranked on a 4-point descriptive scale
Compare blood inflammatory markers between the ARINA-1 and placebo arms | 56 days
  C-reactive protein
Compare changes in mucolytic use between ARINA-1 and placebo arms | 56 days
  Compare the initiation or changes to regimen for drugs such as n-acetylcysteine, dornase alfa, etc. This information will be collected at all clinic visits and phone calls.
Compare changes in airway clearance techniques between ARINA-1 and placebo arms | 56 days
  Compare the initiation or changes to regimen for airway clearance techniques such as chest physical therapy, high-frequency oscillating vest therapy, etc. This information will be collected at all clinic visits and phone calls.
Compare FEV1 between the ARINA-1 and treatment arms | 56 days
  measured in L
Compare FVC between the ARINA-1 and treatment arms | 56 days
  measured in L
Compare FEF25-75 between the ARINA-1 and treatment arms | 56 days
  measured in L/sec
Compare PEF between the ARINA-1 and treatment arms | 56 days
  measured in L/min
Compare sputum percent solids between the ARINA-1 and placebo arms | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Daley, MD, Principal Investigator — National Jewish Health
Locations (10):
- United States (10):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - National Jewish Hospital, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Louisiana State University, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas - Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No